CLINICAL TRIAL: NCT03473197
Title: A 6-Week, Randomized Study to Evaluate the Potential of CCP-020 (Diacerein 1%) Topical Ointment to Induce a Photoallergic Skin Reaction in Healthy Subjects, Using a Controlled Photopatch Test Design
Brief Title: A 6-Week Study to Evaluate the Photoallergic Potential of Diacerein 1% Ointment in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Castle Creek Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CCP-020-105
Record Dates: First submitted 2018-03-05; First posted 2018-03-22 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Healthy
MeSH Terms: interventions — diacerein; Ointments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Cohort (Healthy Volunteers) (Other): Diacerein 1% topical ointment Intra-subject photoallergy (photosensitization) test
  Interventions: Drug: Diacerein 1% ointment

INTERVENTIONS:
Drug: Diacerein 1% ointment — During the 3-week Induction Phase, diacerein 1% ointment and vehicle ointment were applied under fully occlusive patch conditions to two randomly assigned skin sites on the infrascapular region of the back twice each week for approximately 24 hours (±4 hours). After patch removal, one application site and an untreated control site was irradiated, and all sites were evaluated 24 hours, 48 hours, and 72 hours later. Following a rest period, during the Challenge Phase, the study products were applied to two naive sites once for approximately 24 hours (±4 hours). After patch removal, one application site and an untreated control site was irradiated, and all sites were evaluated 24 hours, 48 hours, and 72 hours later. A Re-Challenge was to be performed if a response observed during the Challenge Phase indicated photosensitization.
  Other Names: CCP-020

SUMMARY:
A study in healthy male and female adult volunteers to determine the potential of diacerein 1% ointment to induce a photoallergic skin reaction using a controlled photopatch testing procedure.

DETAILED DESCRIPTION:
This was a randomized, single center, vehicle controlled, within-subject comparison study of diacerein 1% ointment and vehicle ointment applied under fully occlusive patch conditions on the infrascapular region of each subject's back to induce a photoallergic skin reaction following Ultraviolet (UV) irradiation. This was repeated twice each week during the 3-week Induction Phase, once during rest week 4 as applicable and once at Challenge Phase.

ELIGIBILITY:
Key Inclusion Criteria:

* Is a healthy male or female (to be confirmed by medical history);
* Is 18 years of age or older;
* In the case of a female of childbearing potential, is using an acceptable form of birth control;
* In the case of a female of childbearing potential, has a negative urine pregnancy test (UPT) at Day 1 and are willing to submit to a UPT at the end of study (EOS);
* Is free of any systemic or dermatological disorder, which, in the opinion of the Investigator, will interfere with the study results or increase the risk of AEs;
* Is of any Fitzpatrick Skin Type or race, providing the skin pigmentation will allow discernment of erythema

Key Exclusion Criteria:

* Has a history of photosensitivity or photoallergy;
* Is using systemic/topical corticosteroids within 3 weeks prior to and/or during the study, or systemic/topical antihistamines 72 hours prior to and during the study;
* Is not willing to refrain from using systemic/topical anti-inflammatory analgesics such as aspirin, (occasional use of acetaminophen will be permitted);
* Are taking medication known to cause phototoxic reactions (eg, tetracyclines, thiazides, nonsteroidal anti-inflammatory drugs [NSAIDS]);
* Is using medication which, in the opinion of the Investigator, will interfere with the study results;
* Is unwilling or unable to refrain from the use of sunscreens, cosmetics, creams, ointments, lotions or similar products on the back during the study;
* Has psoriasis and/or active atopic dermatitis/eczema;
* Had a known sensitivity or allergy to constituents of the materials being evaluated including diacerein, mineral oil, petrolatum, cetyl alcohol, D&C Yellow #10 and/or ethyl paraben;
* Has damaged skin in or around the test sites, including sunburn, excessively deep tans, uneven skin tones, tattoos, scars, excessive hair, numerous freckles, or other disfigurations of the test site;
* Has received treatment for any type of internal cancer within 5 years prior to study entry;
* Has any known sensitivity to adhesives; and/or
* Has received any investigational drugs(s) with 4 weeks prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Spellman, MD, Study Chair — Castle Creek Pharmaceuticals, LLC
Locations (1):
- TKL Research, Fair Lawn, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Skin sites
Groups:
- Single Cohort (Healthy Volunteers): During the 3-week Induction Phase, diacerein 1% ointment and vehicle ointment were applied under fully occlusive patch conditions to two randomly assigned skin sites on the infrascapular region of the back twice each week for approximately 24 hours (±4 hours). After patch removal, one application site and an untreated control site was irradiated, and all sites were evaluated 24 hours, 48 hours, and 72 hours later. Following a rest period, during the Challenge Phase, the study products were applied to two naive sites once for approximately 24 hours (±4 hours). After patch removal, one application site and an untreated control site was irradiated, and all sites were evaluated 24 hours, 48 hours, and 72 hours later. A Re-Challenge was to be performed if a response observed during the Challenge Phase indicated photosensitization.
Period: Overall Study
Arm/Group | Single Cohort (Healthy Volunteers)
Started | 61; 255 Skin sites
Diacerein 1% Ointment Irradiated | 51; 51 Skin sites
Vehicle Ointment Irradiated | 51; 51 Skin sites
Diacerein 1% Ointment Non-irradiated | 51; 51 Skin sites
Vehicle Ointment Non-irradiated | 51; 51 Skin sites
Untreated Irradiated | 51; 51 Skin sites
Completed | 51; 255 Skin sites
Not Completed | 10; 0 Skin sites
Not completed — Adverse Event | 4
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | Single Cohort (Healthy Volunteers)
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (14.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 54
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 61
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 61

OUTCOME MEASURES:

1. Primary Outcome: Observed Photoallergy (Photosensitization): Number of Skin Sites by Maximum Total Irritation Score
Description: The determination of photosensitization reactions was summarized by frequency counts of the total dermal irritation score during the Challenge Phase. Total Irritation Score is a visual score summing the degree of erythema and edema. Minimum score=0, maximum score=5; higher score=worse outcome
Time Frame: Skin sites evaluated 24, 48, and 72 hours after patch removal and irradiation challenge
Population: The evaluation of photoallergy was based on all subjects who completed the Challenge Phase of the study.
Measure: Number; unit: Number of affected skin sites
Units Other Than Participants: skin sites
Arm/Group | Single Cohort (Healthy Volunteers)
Number analyzed (Participants) | 51
Number analyzed (skin sites) | 255
Number of affected skin sites
  Diacerein irradiated max score 1 at 24 hrs: number analyzed (skin sites) | 51
  Diacerein irradiated max score 1 at 24 hrs | 10
  Diacerein irradiated max score 1 at 48 hrs: number analyzed (skin sites) | 51
  Diacerein irradiated max score 1 at 48 hrs | 3
  Diacerein irradiated max score 1 at 72 hrs: number analyzed (skin sites) | 51
  Diacerein irradiated max score 1 at 72 hrs | 1
  Diacerein non-irradiated max score 1 at 24 hrs: number analyzed (skin sites) | 51
  Diacerein non-irradiated max score 1 at 24 hrs | 0
  Diacerein non-irradiated max score 1 at 48 hrs: number analyzed (skin sites) | 51
  Diacerein non-irradiated max score 1 at 48 hrs | 0
  Diacerein non-irradiated max score 1 at 72 hrs: number analyzed (skin sites) | 51
  Diacerein non-irradiated max score 1 at 72 hrs | 0
  Vehicle irradiated max score 1 at 24 hrs: number analyzed (skin sites) | 51
  Vehicle irradiated max score 1 at 24 hrs | 10
  Vehicle irradiated max score 1 at 48 hrs: number analyzed (skin sites) | 51
  Vehicle irradiated max score 1 at 48 hrs | 3
  Vehicle irradiated max score 1 at 72 hrs: number analyzed (skin sites) | 51
  Vehicle irradiated max score 1 at 72 hrs | 1
  Vehicle non-irradiated max score 1 at 24 hrs: number analyzed (skin sites) | 51
  Vehicle non-irradiated max score 1 at 24 hrs | 0
  Vehicle non-irradiated max score 1 at 48 hrs: number analyzed (skin sites) | 51
  Vehicle non-irradiated max score 1 at 48 hrs | 0
  Vehicle non-irradiated max score 1 at 72 hrs: number analyzed (skin sites) | 51
  Vehicle non-irradiated max score 1 at 72 hrs | 0
  Untreated irradiated max score 1 at 24 hrs: number analyzed (skin sites) | 51
  Untreated irradiated max score 1 at 24 hrs | 16
  Untreated irradiated max score 1 at 48 hrs: number analyzed (skin sites) | 51
  Untreated irradiated max score 1 at 48 hrs | 5
  Untreated irradiated max score 1 at 72 hrs: number analyzed (skin sites) | 51
  Untreated irradiated max score 1 at 72 hrs | 1

ADVERSE EVENTS:
Time Frame: 6 weeks: 3 weeks Induction Period, 2.5 week Rest Period, 0.5 week Challenge Period
Description: Adverse events were not assessed at a patch site specific level.
Arm/Group | Single Cohort (Healthy Volunteers)
All-Cause Mortality (participants affected / at risk) | 0/61
Serious Adverse Events (participants affected / at risk) | 0/61
Other Adverse Events (participants affected / at risk) | 0/61

LIMITATIONS AND CAVEATS:
no limitations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-25): https://cdn.clinicaltrials.gov/large-docs/97/NCT03473197/Prot_SAP_000.pdf